CLINICAL TRIAL: NCT02982421
Title: The Effect of Group Art Therapy on Physical and Psychological Symptoms of Breast Cancer Survivors Receiving Hormonal Therapy
Brief Title: The Effect of Art Therapy on Physical and Psychological Symptoms of Breast Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0304-16-RMC
Record Dates: First submitted 2016-07-24; First posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Research (Experimental): Group Art Therapy
  Interventions: Behavioral: Group art therapy
- Control (Sham Comparator): Participants will receive Psychoeducational material in the form of a lecture and will engage in the coloring of mandalas.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Group art therapy — Participants will engage in an art therapy group tailored at emotion expression related to the experience of breast cancer survivorship.
  Arms: Research
Behavioral: Control — Participants will receive Psychoeducational material in the form of a lecture and will engage in the coloring of mandalas.
  Arms: Control

SUMMARY:
Art Therapy is a health profession in which art making is utilized as a means of expression and communication within a therapeutic and supportive relationship [1]. Art therapy has been shown to reduce psychological (anxiety, negative mood) and physical (pain, fatigue) symptoms which accompany many breast cancer patients and survivors [2-7]. Qualitative studies provide an initial understanding of the mechanisms through which art therapy facilitates symptom reduction [8]. Breast cancer patients have reported that art therapy provided them with access to emotional material otherwise inaccessible [9]. The goal of this study is to examine the effect of art making within a therapeutic framework on emotional awareness and acceptance.

ELIGIBILITY:
Inclusion Criteria:

Adult women (over age 18), breast cancer survivors without evidence of active illness, hebrew speaking and receiving preventative hormonal therapy for at least 6 months (steady state), receiving care at the survivor's clinic of Davidoff Medical Center

Exclusion Criteria:

A psychiatric diagnosis requiring medication, functional difficulties that affect the ability to handle art supplies, non-hebrew speaking, unwilling to answer the research questionnaires

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-05 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Quality of Life: The FACT-B (Hahn et al, 2015) | Change from study start to end of intervention (8 weeks)
  36 item scale

SECONDARY OUTCOMES:
The levels of Emotional Awareness Scale (LEAS; Lane et al, 1990) | Change from study start to end of intervention (8 weeks)
  20 item scale
Acceptance of Emotion Scale (AE; Weihs et al, 2008) | Change from study start to end of intervention (8 weeks)
  13 item scale
Emotional Approach Coping scales (Stanton et al., 2000) | Change from study start to end of intervention (8 weeks)
  36 item scale
The Mindful Attention Awareness Scale (MAAS)(Carlson & Brown, 2005). | Change from study start to end of intervention (8 weeks)
  15 item scale
Center for Epidemiologic Studies Depression Scale (CES-D) (Cohen, 1997) | Change from study start to end of intervention (8 weeks)
  20 item scale
The Generalized Anxiety Disorder scale (GAD-7) (Spitzer, Kroenke, Williams, & Löwe, 2006) | Change from study start to end of intervention (8 weeks)
  7 item scale
The Breast Cancer Prevention Trial (BCPT) Symptom Scales (Stanton et al., 2005) | Change from study start to end of intervention (8 weeks)
  23 item scale

CONTACTS AND LOCATIONS:
Overall Officials: Rinat Yerushalmi, MD, Study Director — Oncology Department, RMC; Tal Granot, MA, RN, Study Director — Davidoff Cancer Center, RMC; Noga Sela, BA, RN, Study Chair — Oncology, RMC; Sylvia Drier, MA, RN, Study Director — Davidoff Cancer Center, RMC
Locations (1):
- Rabin Medical center, Petah Tikva, Israel, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uttley L, Stevenson M, Scope A, Rawdin A, Sutton A. The clinical and cost effectiveness of group art therapy for people with non-psychotic mental health disorders: a systematic review and cost-effectiveness analysis. BMC Psychiatry. 2015 Jul 7;15:151. doi: 10.1186/s12888-015-0528-4. PMID 26149275
- [Background] Archer S, Buxton S, Sheffield D. The effect of creative psychological interventions on psychological outcomes for adult cancer patients: a systematic review of randomised controlled trials. Psychooncology. 2015 Jan;24(1):1-10. doi: 10.1002/pon.3607. Epub 2014 Jun 21. PMID 24953449
- [Background] Monti DA, Peterson C, Kunkel EJ, Hauck WW, Pequignot E, Rhodes L, Brainard GC. A randomized, controlled trial of mindfulness-based art therapy (MBAT) for women with cancer. Psychooncology. 2006 May;15(5):363-73. doi: 10.1002/pon.988. PMID 16288447
- [Background] Nainis N, Paice JA, Ratner J, Wirth JH, Lai J, Shott S. Relieving symptoms in cancer: innovative use of art therapy. J Pain Symptom Manage. 2006 Feb;31(2):162-9. doi: 10.1016/j.jpainsymman.2005.07.006. PMID 16488349
- [Background] Oster I, Svensk AC, Magnusson E, Thyme KE, Sjodin M, Astrom S, Lindh J. Art therapy improves coping resources: a randomized, controlled study among women with breast cancer. Palliat Support Care. 2006 Mar;4(1):57-64. doi: 10.1017/s147895150606007x. PMID 16889324
- [Background] Svensk AC, Oster I, Thyme KE, Magnusson E, Sjodin M, Eisemann M, Astrom S, Lindh J. Art therapy improves experienced quality of life among women undergoing treatment for breast cancer: a randomized controlled study. Eur J Cancer Care (Engl). 2009 Jan;18(1):69-77. doi: 10.1111/j.1365-2354.2008.00952.x. PMID 19473224
- [Background] Thyme KE, Sundin EC, Wiberg B, Oster I, Astrom S, Lindh J. Individual brief art therapy can be helpful for women with breast cancer: a randomized controlled clinical study. Palliat Support Care. 2009 Mar;7(1):87-95. doi: 10.1017/S147895150900011X. PMID 19619378
- [Background] Boehm K, Cramer H, Staroszynski T, Ostermann T. Arts therapies for anxiety, depression, and quality of life in breast cancer patients: a systematic review and meta-analysis. Evid Based Complement Alternat Med. 2014;2014:103297. doi: 10.1155/2014/103297. Epub 2014 Feb 26. PMID 24817896
- [Background] Collie K, Bottorff JL, Long BC. A narrative view of art therapy and art making by women with breast cancer. J Health Psychol. 2006 Sep;11(5):761-75. doi: 10.1177/1359105306066632. PMID 16908471